CLINICAL TRIAL: NCT07384624
Title: Curing HIV: Proof of Concept Randomized Clinical Trial With Pyrimethamine, Lenalidomide, TOpiramate
Brief Title: Combining Latency Reversing Agents to Address the HIV Reservoir
Acronym: PLUTO
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Casper Rokx, Erasmus MC internist-infectious diseases specialist, principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2026-525211-14-00.; 2026-525211-14-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-08; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: HIV (Human Immunodeficiency Virus); HIV -1 Infection
Keywords: HIV; HIV reservoir; Latency Reversing Agent; HIV cure; Topiramate; Pyrimethamine; Lenalidomide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Pyrimethamine; Lenalidomide; Topiramate; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Proof of concept two-phase sequential randomized controlled trial Phase I consists 3 arms of a single dose combination treatment, with a 7-day follow-up.
  Phase II consists of a single arm four-week treatment, with a total follow-up duration of five weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PYR + LENA (Experimental): Pyrimethamine 200mg oral administration + Lenalidomide 25mg oral administration
  Interventions: Drug: Pyrimethamine (PYR); Drug: Lenalidomide
- PYR + TOPI (Experimental): Pyrimethamine 200mg oral administration + Topiramate 400mg oral administration
  Interventions: Drug: Pyrimethamine (PYR); Drug: Topiramate (drug)
- LENA + TOPI (Experimental): Lenalidomide 25mg oral administration + Topiramate 400 mg oral administration
  Interventions: Drug: Lenalidomide; Drug: Topiramate (drug)

INTERVENTIONS:
Drug: Pyrimethamine (PYR) — Pyrimethamine is a registered antiprotozoal agent, which is used for treating toxoplasmosis and malaria. As a latency reversing agent it exerts its effect by targeting the BAF chromatin remodeling complex involved in maintaining a transcriptional repression.
  Arms: PYR + LENA; PYR + TOPI
Drug: Lenalidomide — Lenalidomide is a registered immunomodulatory drug, registered for multipel myeloma, lymphoma's and Kaposi Sarcoma. As an LRA it targets transcription factor IKZF1, a transcriptional repressor.
  Arms: LENA + TOPI; PYR + LENA
Drug: Topiramate (drug) — Topiramate is a drug registered to for migraine prophylaxis and epilepsy. It binds to GRIK5 at the proviral promotor and inhibits its function. GRIK5 derepresses virus transcription initiation with latency reversal as a result.
  Arms: LENA + TOPI; PYR + TOPI

SUMMARY:
The PLUTO trial aims to contribute to the worldwide search for a functional cure of HIV. One the strategies ("shock and kill' strategy) aims to reverse the HIV-reservoir from latency by increasing cell-associated HIV-RNA, which will lead to increased antigen presentation, trigger immune recognition, and facilitate the elimination of reservoir cells. Participants of the trial are adults with HIV with undetectable viral load that are able to give informed consent to participate in the trial, in total 30 patients will be recruited. The investigational medical compounds in this trial are topiramate, lenalidomide and pyrimethamine, which will be combined. These are all licensed drugs for other conditions.

The study consists of two phases. In phase I participants will receive a single dose of the IMPs, as combination therapy. Sampling will be performed before, during and after medical treatment to evaluate latency reversal and safety endpoints. In phase II, participants will receive the combination of IMPs which is the most potent and within safety limits selected from phase I during a four-week treatment. Sampling will take place on a weekly basis to assess latency reversal, reservoir reduction and safety.

Participants will be recruited from the Erasmus MC, Amsterdam university Medical Center, Radboud University Medical Center and the University Medical Center Utrecht.

DETAILED DESCRIPTION:
Rationale Though combined antiretroviral therapy (ART) has made HIV a clinically manageable chronic illness by preventing viral replication, HIV poses great burdens on PLWH and society to this day. Due to the presence of a stable, latent viral reservoir, the virus rebounds when ART is stopped. Additionally this reservoir fuels inflammation with related comorbidities. Finding therapies to reduce the reservoir are therefore an important research objective. One strategy to shrink or eliminate the latent reservoir aims to reverse the reservoir from latency, leading to increased antigen presentation and trigger immune recognition (the "shock and kill" strategy). Several latency reversal agents (LRA) have been identified. Though single LRA treatment are effective to a limited extent, they have not resulted in significant HIV reservoir reduction. PLUTO, aims to study novel combinations of promising LRAs with different targets to reactivate and reduce the latent viral reservoir by identifying the combination with strongest latency reversal of phase I of our study and assessing latency reversal and reservoir decay after prolonged treatment in phase II of our study.

Objectives

Primary objectives phase I:

- To assess the efficacy of LRA combinations during a one day treatment on HIV reservoir reactivation in people living with HIV.

Primary objectives phase II:

- Efficacy of dual LRA combination treatments on HIV reservoir reduction.

Main trial endpoints

Phase I Primary endpoint:

• Fold change in cell-associated HIV-RNA at time points 6, and 24 hours compared to baseline

Phase II Primary endpoint:

• Log transformed HIV-DNA at T=4w compared to T=0

Trial design Proof of concept two-phase sequential randomized controlled trial. Phase I consists of three arms receiving a single dose combination treatment, with a 7-day follow-up.

Phase II consists of a single arm receiving a four-week treatment with the selected treatment from phase I, and a with a total follow-up duration of five weeks.

Trial population Phase I 30 people with HIV-1 with inclusion criteria: ≥18years of age, plasma HIV-RNA >1000c/mL before ART, current plasma HIV-RNA <50c/ml for at least two measurements on uninterrupted ART and current CD4+T-cells > 200/mm3.

Phase II A minimum of 16 people with HIV-1 with the same inclusion criteria. All participants from phase I are eligible, and may move on to, phase II with additional consent. In case the required number of participants are not reached from phase I, new participants can be recruited following the same selection procedure as in phase I.

Interventions Phase I The investigational drugs are Pyrimethamine, Lenalidomide, and Topiramate. Patients will be randomized 1:1:1 in one of three arms to receive a single dose of LRA combination of two investigational drugs

Phase II Compound combination with highest latency reversing potential, within safety limits and taking patient participant preference into account is the phase II intervention. Dosing is adjusted to achieve steady state concentrations similar to phase I.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection, confirmed by 4th generation ELISA, Western Blot or PCR.
* Age ≥ 18 years old.
* Confirmed HIV1, subtype A, B, C or D.
* Uninterrupted ART therapy for a minimum 6 months. .
* Plasma HIV RNA <≤50 copies/ml prior to inclusion at two consecutive measurements at least three months apart.
* No disclosed missed ART on more than 2 days per month.
* Current blood CD4+T-cell count of ≥200 cells/mm3
* No clinical signs of cellular immunodeficiency or AIDS.
* Pre-ART plasma HIV RNA ≥1000 copies/mL.
* Able to understand provided information and to give informed consent.

Exclusion Criteria:

* Prior exposure to any of the studied LRAs in the previous 90 days
* HIV-2 (double)infection
* Co-infection with hepatitis B, unless resolved HBV (anti-HBc positive, anti-HBs positive and HBsAg negative) OR HBsAg positive and on continuous HBV-active antiviral therapy for ≥24 weeks prior to dosing, and HBV DNA undetectable or ≤ 200 IU/mL on two measurements (screening and within 4 weeks prior to enrolment), and no history of advanced fibrosis/cirrhosis (stage F2 and higher)
* Co-infection with hepatitis C, measured by the presence of hepatitis C virus RNA in blood.
* Co-medication with clinically significant interactions with LRA
* mRNA vaccine or adjuvant vaccine (e.g. Shingrix) in the previous 8 weeks.
* Megaloblastic anaemia due to folate deficiency and untreated haemolysis of any cause
* Active malignancy during the past year with the exception of basal carcinoma of the skin, stage 0 cervical carcinoma, Kaposi's sarcoma treated with ART alone or other indolent malignancies.
* History of suicide attempt or suicidal ideation.
* History of ophthalmological medical problems leading to glaucoma or visual field disturbances (e.g. macula oedema). Refraction abnormalities that can be corrected by lenses are acceptable.
* History of any medical condition with a causal relationship with hyperammonemia.
* History of epileptic seizures in the previous year.
* Registered allergies for any of the investigational medical products
* Sexually active participants who do not fit any of the following:

  a) Female subject of childbearing potential willing to comply with pregnancy tests before start and four weeks after end of treatment and willing to use of double contraceptive measures during and until 1 week after administration of study medication. Non-childbearing is defined by one of the following criteria: amenorrhoea for ≥ 1 year, premature ovarian failure, assigned male at birth, or having undergone bilateral salpingo-oophorectomy, or hysterectomy. b) Sexually active male PLWH who have sex with female partners of childbearing potential and willing to abstain from sex or willing to use condom protection during and until 1 week after administration of study medication.

  c) Sexually active male PLWH who have sex with postmenopausal female partners and willing to abstain from sex or willing to use condom protection or with a postmenopausal female partner on pre-exposure prophylaxis during and until 1 week after administration of study medication.

  d) Male PLWH who have sex with male partners and willing to abstain from sex or willing to use a condom protection during and until 1 week after administration of study medication.

  e) Male PLWH who have sex with male partners on preexposure prophylaxis during and until 1 week after administration of study medication.
* Any lab abnormalities at screening as listed below:

  1. Moderate kidney impairment, defined as eGFR <50 mL/min. In PLWH on dolutegravir- or bictegravir-based ART regimens, cystatin C-based eGFR can be used, since possible drug interference with tubular creatinine excretion which leads to eGFR underestimation.
  2. Moderate hepatic impairment, defined as bilirubin > 3 x upper limit of normal (ULN) or ALT > 3x ULN
  3. Inadequate blood counts, defined as: haemoglobin <6.5 mmol/L (males) or <6.0 mmol/L (females), Absolute neutrophil count <1000 cells/mm3, thrombocytes <100 x109/L, international standardized ratio >1.6, activated partial thromboplastin time >40 seconds,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Phase I primary outcome: Fold change in cell-associated HIV-RNA | At time points 6 and 24 hours after treatment, compared to baseline
  The fold change in cell-associated HIV-RNA within and between the study arms
Phase II primary outcome: Log transformed HIV-DNA | At time point 4 weeks compared to baseline
  The change in log transformed HIV-DNA within the treatment group. Measured using IPDA and SQuHIVLa

SECONDARY OUTCOMES:
Phase I & II: Clinical safety and tolerability of the LRA drug combination. | Phase I: 1 week Phase II: 5 weeks
  The number and severity of clinical and biochemical adverse events assessed using Common Terminology Criteria for Adverse Events version 6
Phase I: Participant preference on the latency reversing agent (LRA) combinations. | At 0 hours, 24 hours and 7 days
  Participant preference for LRA combinations, quantitatively assessed using a pill diary with Likert scales 1-5 (higher scores meaning better outcome)
Phase I: Participant quality of life during combination LRA treatment | Baseline, and at timepoint 7 days
  To evaluate qualitative patient reported outcomes of quality of life assessed by semi-structured interviews
Phase I: Plasma HIV-RNA kinetics during interventional treatment | At time points 6 hours, 24 hours and 7 days compared to baseline
  Change in plasma HIV-RNA between and within arms
Phase I: Change of the functionality of immune cells | At 7 days, compared to baseline
  The change of the functionality of innate and adaptive immune cell subpopulations, specifically total T cells and HIV specific CD4+ and CD8+ T cells as well as HIV specific antibody profiles, between and within the groups
Phase I: Change of the phenotype of immune cells | At 7 days, compared to baseline
  The change of the phenotype of innate and adaptive immune cell subpopulations, specifically total T cells and HIV specific CD4+ and CD8+ T cells as well as HIV specific antibody profiles, between and within the groups
Phase I: Pharmacokinetics of LRA compounds | At time points 2 hours, 6 hours, 24 hours and 7 days compared to baseline
  Plasmaconcentrations Cmax will be measured using validated methods and related to the primary endpoint
Phase I: Pharmacokinetics of LRA compounds | At time points 2 hours, 6 hours, 24 hours and 7 days compared to baseline
  Plasmaconcentrations Cthrough will be measured using validated methods and related to the primary endpoint
Phase I: Drug plasma levels of ART | At time points 0 hours, 6 hours, 24 hours and 7 days
  Plasma concentrations Cmax of ART (antiretroviral therapy) will be measured using validated methods and related to LRA compounds
Phase I: Drug plasma levels of ART | At baseline and at time points 6 hours, 24 hours and 7 days
  Description: Plasma concentrations Cthrough of ART (antiretroviral therapy) will be measured using validated methods and related to LRA compounds
Phase I: Ex vivo/ In vivo correlation of reservoir reactivation | From time points baseline to 24 hours
  The correlation between ex vivo and in vivo fold change in cell-associated HIV-RNA
Phase II: Participant quality of life during LRA combination treatment. | At baseline and timepoint 4 weeks
  To evaluate qualitative patient reported outcomes of quality of life assessed by semi-structured interviews
Phase II: Plasma HIV-RNA kinetics during interventional treatment | At timepoints 24 hours, 1 week, 2 weeks, 3 weeks and 4 weeks compared to baseline
  Change in plasma HIV-RNA absolute copies/mL within groups
Phase II: functionality of innate and adaptive immune cells | At time points 1 week, 2 weeks, 3 weeks and 4 weeks compared to baseline
  The change of the functionality of innate and adaptive immune cell subpopulations, specifically total T cells and HIV specific CD4+ and CD8+ T cells as well as HIV specific antibody profiles, between and within the groups
Phase II: Phenotype of innate and adaptive immune cells | At time points 1 week, 2 weeks, 3 weeks and 4 weeks compared to baseline
  The change of the phenotype of innate and adaptive immune cell subpopulations, specifically total T cells and HIV specific CD4+ and CD8+ T cells as well as HIV specific antibody
Phase II: Pharmacokinetics LRA compounds | At time points 1 week, 2 weeks, 3 weeks and 4 weeks compared to baseline
  Plasmaconcentrations Cmax will be measured using validated methods and related to the primary endpoint
Phase II: Pharmacokinetics of LRA compounds | At time points 1week, 2 weeks, 3 weeks and 4 weeks compared to baseline
  Plasmaconcentrations Cthrough will be measured using validated methods and related to the primary endpoint
Phase II: Drug plasma levels of ART | At time points 1 week, 2 weeks, 3 weeks and 4 weeks
  Plasma concentrations Cmax of ART will be measured using validated methods. The pharmacokinetic profiles ART will be assessed in relation to the primary endpoint and LRA compounds
Phase II: Drug plasma levels of ART | At time points 1 week, 2 weeks, 3 weeks, 4 weeks
  Description: Plasma concentrations Cthrough of ART will be measured using validated methods. The pharmacokinetic profiles ART will be assessed in relation to the primary endpoint and LRA compounds

OTHER OUTCOMES:
Inflammatory biomarkers during LRA treatment | At time points 24 hours, 1 week and 4 weeks compared to baseline
  Assessment of serum inflammatory biomarkers on LRA treatment
Cellular transcriptomic responses before and after exposure to LRA | At time points 24 hours, 1 week and 4 weeks compared to baseline
  Change in host and HIV-related gene expression profile in CD4+ T-cell reservoir cells by RNA sequencing on pathways of immune modulation and off-target effects within and between groups
Viral reservoir myeloid or lymphoid cell origin | At baseline and time points 24 hours, 1 week and 4 weeks
  Viral envelop myeloid and lymphoid cell tropism by RNA sequencing
Trained immunity during LRA exposure | At time points 24 hours, 1 week and 4 weeks compared to baseline
  Change in transcriptome and epigenetic histone modification in trained monocytes following ex vivo stimulation with several pathogens and ligands of peripheral blood mononuclear cells (PBMC)
Identification of clinical predictors of LRA responses. | Cell associated HIV-RNA from baseline to 24 hours and change in HIV-DNA from baseline to 4 weeks.
  The mean difference in fold change in cell associated HIV-RNA and change in HIV-DNA between HIV related and demographical variables.
Synergy of LRA combination using historic controls on LRA monotherapy | From baseline to 24 hours
  The fold change in cell-associated HIV-RNA on combined LRA treatment compared to each LRA as monotherapy in historic controls from previous randomized clinical trials (LUNA/ORBIT/STAR)

CONTACTS AND LOCATIONS:
Overall Officials: Casper Rokx, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Center, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored under FAIR use principle for use in future research. Should external researchers want to use this dataset, they can contact the principal investigator. In the case of adequate privacy standards data can be shared under a specific new Data Sharing Agreement
Supporting Information: SAP, Analytic Code
Time Frame: Data will be available after publication of primary results. Data will kept in storage for 25 years
Access Criteria: Receiving facility has data privacy protection meeting EU GDPR standards